CLINICAL TRIAL: NCT03142568
Title: Safety of Sildenafil in Premature Infants at Risk of Bronchopulmonary Dysplasia
Brief Title: Safety of Sildenafil in Premature Infants
Acronym: SIL02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-2436; 75N94022F00001 (Other Grant/Funding Number: NICHD); R01FD006099-01 (FDA)
Record Dates: First submitted 2017-04-17; First posted 2017-05-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sildenafil cohort 1 (Experimental): Within cohort 1 infants will be randomized using a 3:1 scheme to receive sildenafil or placebo. Infants randomized to sildenafil will receive 0.125 mg/kg daily every 8 hours intravenously (IV), or 0.25 mg/kg daily every 8 hours enterally for 28 days.
  Interventions: Drug: Sildenafil
- Placebo cohort 1 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent of dextrose 5% (sugar water) to be administered IV or enteral use.
  Interventions: Other: Placebo
- Sildenafil cohort 2 (Experimental): Cohort 2 infants will receive sildenafil 0.5 mg/kg daily every 8 hours intravenously (IV) or 1 mg/kg daily every 8 hours enterally for 28 days.
  Interventions: Drug: Sildenafil
- Placebo cohort 2 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent of dextrose 5% (sugar water) to be administered IV or enteral use.
  Interventions: Other: Placebo
- Sildenafil cohort 3 (Experimental): Cohort 3 infants will receive sildenafil 1 mg/kg daily every 8 hours intravenously (IV) or 2 mg/kg daily every 8 hours enterally for 28 days.
  Interventions: Drug: Sildenafil
- Placebo cohort 3 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent of dextrose 5% (sugar water) to be administered IV or enteral use.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sildenafil — Infants will be randomized using a 3:1 scheme to receive sildenafil or placebo.
  Other Names: Revatio
  Arms: Sildenafil cohort 1; Sildenafil cohort 2; Sildenafil cohort 3
Other: Placebo — Infants randomized to the placebo group will receive the equivalent volume of dextrose 5% for IV use or enteral use (if receiving enteral study drug).
  Other Names: sugar water
  Arms: Placebo cohort 1; Placebo cohort 2; Placebo cohort 3

SUMMARY:
Describe the safety of sildenafil in premature infants at risk of bronchopulmonary dysplasia and determine preliminary effectiveness and pharmacokinetics (PK) of sildenafil. Funding Source - FDA OOPD.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, placebo-controlled, sequential dose escalating, double masked, safety data study of sildenafil in premature infants.

This is a Phase II study design, premature infants (inpatient in neonatal intensive care units) will be randomized in a dose escalating approach 3:1 (sildenafil: placebo) into 3 cohorts with escalating doses of sildenafil. There will be 40 randomized and dosed participants in each cohort for a total of up to 120 participants. Cohort 1 sildenafil dose will be 0.125 mg/kg q 8 hours IV or 0.25 mg/kg q 8 hours enteral. Cohort 2 sildenafil dose will be 0.5 mg/kg q 8 hours IV or 1.0 mg/kg q 8 hours enteral. Cohort 3 sildenafil dose will be 1 mg/kg q 8 hours IV or 2 mg/kg q 8 hours enteral.

ELIGIBILITY:
Inclusion Criteria:

* Receiving positive airway pressure (nasal continuous airway pressure, nasal intermittent positive pressure ventilation, or nasal cannula flow > 1LPM) or mechanical ventilation (high frequency or conventional)
* <29 weeks gestational age at birth
* 7-28 (inclusive) days postnatal age at time of randomization

Exclusion Criteria:

* Currently receiving vasopressors
* Currently receiving inhaled nitric oxide
* Baseline mean arterial pressure < gestational age (in weeks) plus postnatal age (in weeks) within 2 hours of sildenafil administration
* Known allergy to sildenafil
* Known sickle cell disease
* AST > 225 U/L < 72 hours prior to randomization
* ALT > 150 U/L < 72 hours prior to randomization

Ages: 7 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Safety as determined by adverse event experienced by participants | 42 days for each participant
  Description of safety of sildenafil in premature infants at risk of BDP. Safety will be assessed following initial study-specific procedure e.g., screening blood draws, dosing through 14 days post last study dose and it will be assessed by frequency and incidence of adverse events and serious adverse events.

SECONDARY OUTCOMES:
Volume of Distribution | Samples collected after any dose following completion of 14 days of study drug administration.
  Volume of distribution [ Time Frame: 8 hr. dosing: time frame: 0-15 min, 30-60 min, 1-2, 2-3, 3-4, 4-5, within 15 min prior to next dose, and 16-24 hrs. after last dose.]
Clearance | Samples collected after any dose following completion of 14 days of study drug administration.
  Clearance [ Time Frame:8hr dosing: time frame: 0-15 min, 30-60 min, 1-2, 2-3, 3-4, 4-5, within 15 min prior to next dose, and 16-24 hrs. after last dose.]
Half-Life | Samples collected after any dose following completion of 14 days of study drug administration.
  Half-life [ Time Frame: 8hr. dosing: time frame: 0-15 min, 30-60 min, 1-2, 2-3, 3-4, 4-5, within 15 min prior to next dose, and 16-24 hrs. after last dose.
Area Under the Curve (AUC) | Samples collected after any dose following completion of 14 days of study drug administration.
  Area under the plasma concentration versus time curve (AUC) of sildenafil. [Time Frame: 8hr. dosing: time frame: 0-15 min, 30-60 min, 1-2, 2-3, 3-4, 4-5, within 15 min prior to next dose, and 16-24 hrs. after last dose.]
Peak Plasma Concentration | Samples collected after any dose following completion of 14 days of study drug administration.
  Maximum concentration Peak Plasma Concentration (Cmax) of sildenafil [Time Frame: 8hr. dosing: time frame: 0-15 min, 30-60 min, 1-2, 2-3, 3-4, 4-5, within 15 min prior to next dose, and 16-24 hrs. after last dose.]
Change in moderate-severe BPD or death risk from baseline | 36 weeks postmenstrual age
  Moderate-severe BPD or death risk will be defined by the NICHD Neonatal Research Network BPD outcome estimator. https://neonatal.rti.org/
  The BPD outcome estimator uses the following information to provide individual risk of BPD:
  1. Gestational age (weeks)
  2. Birth weight (g)
  3. Sex
  4. Maternal Race/Ethnicity
  5. Postnatal day
  6. Ventilation type (on the postnatal day of interest)
  7. FiO2 (%) (on the postnatal day of interest)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Laughon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (15):
- United States (14):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Florida College of Medicine Jacksonville-Wolfson Children's Hospital, Jacksonville, Florida
  - University of Florida Jacksonville Shands Medical Center, Jacksonville, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Hospital of Nevada at UMC, Las Vegas, Nevada
  - Monmouth Medical Center, Long Branch, New Jersey
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Golisano Children's Hospital - University of Rochester Medical Center, Rochester, New York
  - WakeMed Health and Hospitals, Raleigh, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
- Health Sciences Centre Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No